CLINICAL TRIAL: NCT03530254
Title: International Multi-center, Randomized and Controlled Clinical Study, to Evaluate the Clinical Benefit of the ERA Test in Infertile Patients Undergoing Assisted Reproduction Treatment and Medical Indication of PGT-A.
Brief Title: Clinical Study of PGT-A Versus PGT-A+ERA
Acronym: PGT-A&ERA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment speed, higher percentage drop-out and SARS-CoV-2 pandemic situation
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IGX1-P&E-DV-17-08
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Infertility of Uterine Origin
Keywords: Endometrial receptivity; Preimplantation Genetic Diagnosis (PGD); Preimplantation Genetic Testing for Aneuploidy (PGT-A); Embryo Transfer (ET); Endometrial Receptivity Analysis (ERA); Endometrial Diagnosis; Live Newborn Rate (LBR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGT-A without ERA (Other): Patients with PGT-A indication and ET in a Hormone Replacement Therapy (HRT cycle) according to the usual clinical practice (day 5 of progesterone supplementation: P+5/120h).
  Interventions: Diagnostic Test: PGT-A
- PGT-A and test ERA (Other): Patients with PGT-A indication and pET in HRT cycle following the ERA test indication (when the WOI is confirmed as "Receptive").
  Interventions: Diagnostic Test: PGT-A; Diagnostic Test: ERA Test

INTERVENTIONS:
Diagnostic Test: PGT-A — PGT-A will be carried out following the usual clinical practice. Trophectoderm biopsy samples from blastocysts are analyzed by NGS to screen for numerical chromosomal abnormalities.
Diagnostic Test: ERA Test — The ERA test requires an endometrial biopsy and will determine if the endometrium is receptive or not by analysing the expression levels of 236 genes involved in endometrial receptivity, to assess the optimal time to place an embryo into the uterus and promote a successful implantation and pregnancy.
  Arms: PGT-A and test ERA

SUMMARY:
Patients who have shown previous implantation failures, despite transferring good quality and chromosomally normal embryos (diagnosed by PGT-A), could have a displaced Window of Implantation (WOI) and consequently, alterations in their endometrial receptivity. The correction of this displacement can improve the results of the Assisted Reproduction Treatments (ART).

The ERA test (Endometrial Receptivity Analysis) evaluates the transcriptomic endometrial profile to determine if the patient's uterus is receptive when the embryo is transferred during an In Vitro Fertilization (IVF) process, and identifies the personalized WOI of the patient. This process is called Personalized Embryo Transfer (pET).

The Preimplantation Genetic Test of Aneuploidies or PGT-A (Preimplantation Genetic Testing for Aneuploidy), is currently carried out using Next Generation Sequencing (NGS) and serves to identify chromosomally normal embryos prior to their transfer in an IVF treatment. Aneuploidies are rarely compatible with life or can cause congenital diseases. So, the identification of chromosomally normal embryos, improves the success of reproduction in cases in which infertility is caused by such aneuploidies.

Therefore, the aim of this study is to determine, in a randomized and prospective way, the clinical benefit of adding the ERA test to the embryonic aneuploidies test for patients with a PGT-A indication.

DETAILED DESCRIPTION:
The lack of receptivity of the uterus and chromosomal abnormalities in the embryo are the two main causes of implantation failure. Patients with implantation failure, should consider the PGT-A test to identify and select euploid embryos. In addition, it should be evaluated the endometrium receptivity state at the time of Embryo Transfer (ET).

The PGT-A is an important genetic test that was developed to select embryos during IVF treatment and avoid embryonic chromosomal abnormalities that lead to miscarriage or life born with chromosomal diseases. Embryonic aneuploidy is linked to maternal age. The most common consequences are implantation failure, miscarriage or life born with multiple congenital anomalies. The transfer of euploid embryos (chromosomally normal) diagnosed by PGT-A has shown an increase in implantation rates.

Morphology is the most traditional and routine method of embryo selection being used. However, it is difficult to distinguish normal and abnormal embryos by observing their morphology under a microscope. Therefore, morphological analysis should not be the only technique used to decide which embryo should be transferred. Application of NGS in PGT-A cycles demonstrates that this methodology is reliable, allowing identification and transfer of euploid embryos resulting in ongoing pregnancies. However, despite the transfer of morphologically normal euploid embryos, it is not always possible to acquire optimal results in Assisted Reproductive Techniques (ART).

On the other hand, the endometrial gene expression profile allows the diagnosis of the endometrium receptivity status. This is carried out by a molecular tool developed and patented by Igenomix (PCT/ES2009/00386). The ERA test is a customized expression microarray that identifies the transcriptomic expression profile signature of the personalized Window of Implantation (pWOI). A bioinformatic predictor determines the moment of maximum receptivity, indicating the best time to perform a pET.

If the result of the ERA test is "Receptive", the WOI and the moment of taking the biopsy overlap. Nevertheless, if the result is "Pre-Receptive", the optimal implantation window is expected to be after the moment in which the biopsy is taken, and if the diagnosis is "Post-Receptive", the optimal window of implantation is prior to the biopsy. In a subsequent cycle, a pET will be performed according to the ERA test results.

Recently, it has been conducted a pilot study in patients with previous implantation failures with PGT-A and euploid embryo transfer (ET). The results of the ERA test have shown that a high percentage of these patients have been diagnosed as Non-receptive (90%). This percentage is higher than the expected in the normal population (12-20%) or in the Repeated Implantation Failure (RIF) patients without PGT-A (25-30%). Once the pET was performed according to the results of the ERA test, the gestation rate was 55.55%.

So, the objective of the present study is to validate these preliminary results in a prospective, multi-center, randomized and controlled study to demonstrate the value of the endometrial factor and the improvement of the results obtained in patients with PGT-A indication. If confirmed, it would be recommended the ERA test for all ART patients, not only for those with PGT-A, demonstrating the significance in searching for the pWOI to improve reproductive outcomes.

Considering a maximum drop-out rate of 30%, a total of 750 participants are expected to be included. According to the approved protocol, an interim analysis is planned at 50% of the total enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Majority of age patients whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Patients who already have frozen euploid blastocysts (day 5/6 development) analysed by PGT-A.
* Patients with embryos obtained from their own oocytes fertilized by Intracytoplasmic Sperm Injection (ICSI) or In vitro fertilization (IVF).
* Patients with an expected embryo transfer of one or two embryos (Single ET or Double ET) in a HRT cycle.
* Body Mass Index: 18,5-30 Kg/m2.

Exclusion Criteria:

* Presence of pathologies or malformations that affect the uterine cavity such as polyps, intramural myomas ≥ 4cm or submucosal, septum or hydrosalpinx during the patient's participation in the study. Patients suffering these pathologies before or after their inclusion in the study are allowed to participate if the pathology is corrected before performing any study procedure.
* Any illness or medical condition that is unstable or which, according to medical criteria, may put at risk the patient's safety and her compliance in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Majority of age infertile patients who already have frozen euploids blastocysts (day 5/6 development) obtained from their own oocytes, fertilized by IFV/ICSI and analysed by PGT-A, with an expected embryo transfer of one or two embryos in a Hormone Replacement Therapy cycle (HRT cycle).
Enrollment: 368 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 40 weeks
  Number of babies born per embryo transfer

SECONDARY OUTCOMES:
Implantation rate | 12 weeks
  Number of implanted embryos per total number of embryos transferred
Clinical pregnancy | 20 weeks
  Number of clinical pregnancies per total number of pregnancies
Biochemical pregnancy | 20 weeks
  Number of biochemical pregnancies per total number of pregnancies
Clinical miscarriages | 20 weeks
  Number of clinical miscarriages per total number of pregnancies
Ectopic pregnancies | 20 weeks
  Number of ectopic pregnancies per total number of pregnancies
Obstetric complications | 40 weeks
  Type and number of obstetric complications during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD PhD, Study Chair — Igenomix
Locations (15):
- United States (2):
  - Ovation Fertility Newport Beach, Newport Beach, California
  - Fertility Centers of New England, Reading, Massachusetts
- Pregna Medicina Reproductiva, CABA, Argentina
- Vida Bem Vinda, São Paulo, Brazil
- Olive Fertility Center, Vancouver, Canada
- Shady Grove Fertility Chile, Vitacura, Chile
- Georgian- American Center for Reproductive Medicine ReproART, Tbilisi, Georgia
- India (2):
  - OASIS centre for reproductive medicine, Banjara Hills, Hyderabad
  - Mother And Child Hospital, Defence Colony, National Capital Territory of Delhi
- NASCERE, Mexico City, Mexico City, Mexico
- Spain (2):
  - Milenium Centro Médico y de Bienestar de Alcobendas - Sanitas, Alcobendas, Madrid
  - Instituto Extremeño de Reproducción Asistida S.L. (IERA), Badajoz
- Taiwan IVF Group, Zhubei, Taiwan
- Bahceci Group, Istanbul, Turkey (Türkiye)
- Vinmec Time City International Hospital, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: No